CLINICAL TRIAL: NCT05635695
Title: Assessment of Cultural Pathways in the City Developed on a Smartphone Application on Physical Abilities, Well-being and Sustainable Health Knowledge
Brief Title: Cultural Pathways to Develop Sustainable Health
Acronym: ART'M2-APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Anne-Violette Bruyneel, Professor, School of Health Sciences Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APP-112187
Record Dates: First submitted 2022-11-14; First posted 2022-12-02 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sedentary Behavior
Keywords: Sustainable health; Physical Activity; Cultural pathways; App; Sedentary
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Museum visit (Active Comparator): Free museum visit during 45 to 75 minutes
  Interventions: Other: Free Museum visit
- Cultural pathways App (Experimental): Cultural pathways App during 45 to 75 minutes
  Interventions: Other: Cultural pathways App

INTERVENTIONS:
Other: Free Museum visit — People are tested when they arrive at the museum. Then, they freely visit the different rooms for 45 to 75 minutes. No instructions are given.
  Arms: Free Museum visit
Other: Cultural pathways App — Cultural pathways in the park of the museum will be proposed to people with a smartphone application that will give directions, cultural and sustainable health contents, points of interest with games and specific information about the pathways (distance, noise level, walkability, practical information). There will be two possible levels: contemplative or active.
  Arms: Cultural pathways App

SUMMARY:
The 2030 Agenda for Sustainable Development, adopted by all United Nations Member States in 2015 includes the goal 3 "Ensure healthy lives and promote well-being for all at all ages". One of the essential axes is to promote primary prevention in order to avoid the emergence of diseases and the treatments use with a high environmental impact. Physical activity (PA) is a means of primary prevention known to be very effective in the fight against chronic diseases.

Despite the recommendations on PA, a high number of people are sedentary and in particular in older persons. The main barriers are accessibility and lack of motivation for traditional PA. The investigators believe that the development of cultural pathways could be an excellent way to improve people's health.

The objective of this study is to assess the effects of cultural pathways on the physical abilities, well-being and sustainable health knowledge of sedentary people over 50 years old. This intervention will be compared to a control group visiting a museum freely. The hypothesis is that cultural pathways including games induce enough steps to be considered an effective activity to fight sedentary lifestyle. The number of steps should be higher than the control group. Fatigue, stress and well-being should be improved after the visit as well as sustainable health knowledge.

All the tests will be carried out during the same day by experienced physiotherapists. Physical and well-being tests will be performed before and after the intervention or control. The number of steps taken during the cultural activity will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Sedentary condition (<150 minutes of physical activity per week)
* Medical stability
* Walking independently with or without assistance
* Ability to understand the instructions

Exclusion Criteria:

* Refusal to participate;
* Person with other conditions affecting independent walking;
* Contraindications to prolonged standing;
* Concomitant pathologies that may interfere with the results;
* Inability to follow the study procedure (cognitive disorders, dementia, psychological disorders, language problems...).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Number of steps during cultural activity in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  An activity tracker on the visitor's wrist will measure the number of steps taken while visiting the museum free or with app. Parameter: number of steps.

SECONDARY OUTCOMES:
Change from baseline (pre-visit): fatigue in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  The fatigue will be tested with the Numeric Rating Scale. Parameter: 10-points score (1 = no fatigue, 10 = maximal fatigue).
Change from baseline (pre-visit): stress in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  The stress will be tested with the Numeric Rating Scale. Parameter: 10-points score (1 = no stress, 10 = maximal stress).
Change from baseline (pre-visit): pain in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  The pain will be tested with the Numeric Rating Scale. Parameter: 10-points score (1 = no pain, 10 = maximal pain).
Change from baseline (pre-visit): perceived balance in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  The perceived balance will be tested with a 5-points scale (1 = poor balance ; 5 = excellent balance)
Change from baseline (pre-visit): survey about "sustainable health knowledge" (questionnaire en santé durable in french - QSDFr) in the 2 groups (free visit vs.cultural pathways) | 75 minutes
  The QSDFr will be tested with 8 questions. For each question a score from 0 to 2 will be given (0 = wrong answer, 1 = partial answer, 2 = right answer). The maximal score = 16 points and minimal = 0 points.
Change from baseline (pre-visit): Activities-Specific Balance Confidence (ABC-scale short version) (only intervention group) | 75 minutes
  6-item self-report measure in which individuals rate their balance confidence for performing activities. Items are rated on a rating scale that ranges from 0 (no balance confidence) - 100 (complete balance confidence). Overall score is calculated by adding item scores and then dividing by the total number of items.
Change from baseline (pre-visit): Postural control (only intervention group) center of pressure displacement | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure displacement (mm).
Change from baseline (pre-visit): Postural control (only intervention group) center of pressure velocity | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure velocity (mm/s).
Change from baseline (pre-visit): Postural control (only intervention group) center of pressure sway area | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure sway area (mm2).
Change from baseline (pre-visit): gait speed and dual task (only intervention group) | 75 minutes
  The gait speed will be tested with the Ten-meter walking test in normal walking, fast walking and in dual-task. Parameter: gait speed (m/s)
Change from baseline (pre-visit): museum well-being measures (only intervention group) | 75 minutes
  The well-being will be tested with the museum well-being survey. A generic well-being questionnaire will be used with 12-item version. Each statement is rated out of five depending on the extent of agreement with it (1 = None of the time; 2 = Not very often; 3 = Some of the time; 4 = Very often; 5 = All of the time). The maximal score is 60 points (excellent well-being) and minimal score 12 points (poor well-being).
Change from baseline (pre-visit): museum well-being umbrella measures (only intervention group) | 75 minutes
  The well-being will be tested with the museum well-being umbrella: positive well-being umbrella and negative well-being umbrella. Each of the six sections has a word next to it related to a well-being mood or emotion and numbers from one (I don't feel) to five (I feel extremely). Participants are required to rate the extent they feel the well-being word at that moment in time by circling the appropriate number, following the instructions provided. For both umbrella, maximal score = 30, minimal score = 6.
Safety endpoint: pain (Numeric Rating Scale) | 3 hours
  The safety endpoint will be tested with the pain (Numeric Rating Scale). Parameter: 10-points score (1 = no pain, 10 = maximal pain).
Safety endpoint: fatigue (Numeric Rating Scale) | 3 hours
  The safety endpoint will be tested with the fatigue (Numeric Rating Scale). Parameter: 10-points score (1 = no fatigue, 10 = maximal fatigue).
Safety endpoint: number of subjects who completed the cultural activity and tests. | 3 hours
  The number of subjects who completed the cultural activity and tests will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Violette Bruyneel, Principal Investigator — Geneva School of Health Sciences
Locations (1):
- Geneva School of Health Sciences, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion
Access Criteria: At the end of the project the data will be deposited in the Yareta repository developed by the University of Geneva OR in an institutional repository. This choice will ensure that data is archived and shared in accordance with FAIR principles.

REFERENCES:
- [Background] Harvey JA, Chastin SF, Skelton DA. Prevalence of sedentary behavior in older adults: a systematic review. Int J Environ Res Public Health. 2013 Dec 2;10(12):6645-61. doi: 10.3390/ijerph10126645. PMID 24317382
- [Background] Tudor-Locke C, Craig CL, Aoyagi Y, Bell RC, Croteau KA, De Bourdeaudhuij I, Ewald B, Gardner AW, Hatano Y, Lutes LD, Matsudo SM, Ramirez-Marrero FA, Rogers LQ, Rowe DA, Schmidt MD, Tully MA, Blair SN. How many steps/day are enough? For older adults and special populations. Int J Behav Nutr Phys Act. 2011 Jul 28;8:80. doi: 10.1186/1479-5868-8-80. PMID 21798044
- [Background] Camic PM, Chatterjee HJ. Museums and art galleries as partners for public health interventions. Perspect Public Health. 2013 Jan;133(1):66-71. doi: 10.1177/1757913912468523. PMID 23308010